CLINICAL TRIAL: NCT00116467
Title: Vaccination in the Peripheral Stem Cell Transplant Setting for Acute Myelogenous Leukemia: The Use of Autologous Tumor Cells With an Allogeneic GM-CSF Producing Cell Line
Brief Title: Vaccination in the Peripheral Stem Cell Transplant Setting for Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-0009; K-0009
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML; Acute Myelogenous Leukemia; GVAX; Vaccine; Stem Cell Transplant; Autologous
MeSH Terms: conditions — Leukemia, Myeloid, Acute

INTERVENTIONS:
Biological: GVAX leukemia vaccine (therapeutic cellular vaccine, GM-CSF producing)

SUMMARY:
The purpose of this study is to evaluate clinical and laboratory safety associated with the administration of GVAX leukemia vaccine and to determine the feasibility of generation of GVAX leukemia vaccine in subjects with acute myelogenous leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of de novo AML with no preexisting hematologic dysplasia for more than 3 months.
* No prior therapy except leukapheresis or less than 72 hours of hydroxyurea.

Exclusion Criteria:

* Prior myelodysplastic disorder, or treatment-related leukemia.
* Prior myeloproliferative disease.
* Acute promyelocytic leukemia (APL).
* Prior chemotherapy for a malignant or nonmalignant disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55
Dates: Start 2001-03; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Borrello IM, Levitsky HI, Stock W, Sher D, Qin L, DeAngelo DJ, Alyea EP, Stone RM, Damon LE, Linker CA, Maslyar DJ, Hege KM. Granulocyte-macrophage colony-stimulating factor (GM-CSF)-secreting cellular immunotherapy in combination with autologous stem cell transplantation (ASCT) as postremission therapy for acute myeloid leukemia (AML). Blood. 2009 Aug 27;114(9):1736-45. doi: 10.1182/blood-2009-02-205278. Epub 2009 Jun 25. PMID 19556425